CLINICAL TRIAL: NCT04478383
Title: Repair of Achilles Sleeve Avulsion: a New Transosseous Suture Technique
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018008
Record Dates: First submitted 2020-06-27; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Achilles Tendon Rupture; Fracture, Avulsion
Keywords: Sleeve Avulsion; Achilles Tendinopathy; Suture, transosseous; Achilles Tendon
MeSH Terms: conditions — Fractures, Avulsion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: a new transosseous suture technique — a new technique using the spur base on the insertional site to drill the suture tunnel to repair Achilles sleeve avulsion.

SUMMARY:
This retrospective study identified 12 patients with Achilles sleeve avulsion from November 2013 to March 2016, aiming to explore a new transosseous suture technique for the repair of Achilles sleeve avulsion and observe the short-term curative effect.

DETAILED DESCRIPTION:
Purpose: To explore a new transosseous suture technique for the repair of Achilles sleeve avulsion and observe the short-term curative effect.

Methods:In total, 11 patients diagnosed with Achilles sleeve avulsion underwent this new surgical technique and were followed for a mean time of 40 months. Clinical outcomes were measured using the visual analog scale (VAS), American Orthopaedic Foot & Ankle Society (AOFAS) score, Victorian Institute of Sports Assessment-Achilles (VISA-A) score, Tegner score, and time taken to return to activities. Preoperative and postoperative MRI, the ability to perform heel rise, and complications were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* clinical presentations and physical examination, routine ankle X ray and MRI

Exclusion Criteria:

* calcaneal tuberosity avulsion fractures
* Achilles tendon rerupture
* previous surgical procedure on the affected Achilles tendon

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: One patient was lost to follow-up because she could not be contacted, having moved out of the country. The remaining 11 patients (10 men and one woman, average age: 46 years) were reviewed with an average follow-up time of 40 months (30-57 months).
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
change of Victorian Institute of Sports Assessment-Achilles score | from pre-surgery to two years after surgery
  The VISA-A questionnaire displayed construct validity when used in two populations of patients with Achilles tendinopathy and control subjects. The questionnaire avoids the redundant components of non-specific scoring systems such as that developed for hind foot problems by the American Orthopaedic Society, and those devised for Achilles tendon rupture. Results range from 0 to 100, where 100 represents the perfect score.
change of visual analog scale | from pre-surgery to two years after surgery
  The Visual Analogue Scale (VAS) is designed to present to the respondent a rating scale with minimum constraints. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain they experienced. This gives them the greatest freedom to choose their pain's exact intensity. It also gives the maximum opportunity for each respondent to express a personal response style. The minimum and maximum values of VAS are 10 and 0, respectively. And higher scores mean a worse outcome.
change of American Orthopaedic Foot & Ankle Society score | from pre-surgery to two years after surgery
  The American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Score combines subjective scores of pain and function provided by the patient with objective scores based on the surgeon's physical examination of the patient (to assess sagittal motion, hindfoot motion, ankle-hindfoot stability and alignment of the ankle-hindfoot). The scale includes nine items that can be divided into three subscales (pain, function and alignment). The minimum and maximum values of AOFAS are 100 and 0, respectively. And higher scores mean a better outcome.
change of Tegner score | from pre-surgery to two years after surgery
  The Tegner activity scale was first described in 1985 and initially designed for physician administration after ACL and meniscal injuries. To date, the Tegner activity score has been a frequently used patient-administered activity rating system for patients with various knee disorders. The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Haidian District, China

IPD SHARING:
Plan to Share IPD: No